CLINICAL TRIAL: NCT05560009
Title: Utility of 18F-DOPA PET/MRI Metrics as a Biomarker for Treatment Response Assessment in Sarcoma Patients: A Pilot Study
Brief Title: An Imaging Agent (Fluorodopa F 18) With Positron Emission Tomography/Magnetic Resonance Imaging for Assessing Treatment Response in Patients With High-Grade Soft Tissue Sarcomas
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: MC220702; NCI-2022-04924 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21-005244 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2022-09-19; First posted 2022-09-29 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Recurrent Soft Tissue Sarcoma; Resectable Soft Tissue Sarcoma; Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — fluorodopa F 18; Magnetic Resonance Spectroscopy; Radiotherapy; Radiation; Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (18F-DOPA PET/MRI): Patients receive 18F-DOPA IV and undergo PET/MRI over 60 minutes before standard of care radiotherapy and/or before standard of care surgery.
  Interventions: Drug: Fluorodopa F 18; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Radiation: Radiation Therapy; Procedure: Surgical Procedure

INTERVENTIONS:
Drug: Fluorodopa F 18 — Given IV
  Other Names: (18F)FDOPA; 18F-DOPA; 18F-FDOPA; 3-(2-Fluoro-(sup 18)F-4,5-dihydroxyphenyl)-L-alanine; 6-(18F)Fluoro-L-DOPA; Fluorine F 18 Fluorodopa; Fluorine-18-fluoro-L-DOPA; Fluorodopa (18F); FLUORODOPA F-18; L-6-(18F)Fluoro-DOPA
Procedure: Magnetic Resonance Imaging — Undergo PET/MRI
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Procedure: Positron Emission Tomography — Undergo PET/MRI
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging
Radiation: Radiation Therapy — Receive standard of care radiation therapy
  Other Names: Cancer Radiotherapy; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Procedure: Surgical Procedure — Undergo standard of care surgery
  Other Names: Operation; Surgery; Surgery Type; Surgical; Surgical Intervention; Surgical Interventions; Surgical Procedures; Type of Surgery

SUMMARY:
This study evaluates the use of a new imaging agent called fluorodopa F 18 (18F-DOPA) with positron emission tomography/magnetic resonance imaging (PET/MRI) for assessing treatment response in patients undergoing standard of care radiation therapy and/or surgery for high-grade soft tissue sarcomas that are new or that have come back (recurrent). Though there have been improvements in treatment options for soft tissue sarcomas, there is currently a need for a non-invasive way to determine a patient's potential benefit from receiving one of these treatments. 18F-DOPA with PET/MRI allows a patient's tumor to be visualized and their response to a given treatment assessed.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the correlation between 18F-DOPA PET/MRI quantitative metrics after neoadjuvant treatment (pre-surgery) with percent tumor necrosis.

SECONDARY OBJECTIVE:

I. Compare the changes in 18F-DOPA PET/MRI quantitative metrics between baseline (before radiotherapy [RT]) and after RT, but before surgery with percent tumor necrosis.

OUTLINE:

Patients receive 18F-DOPA intravenously (IV) and undergo PET/MRI over 60 minutes before standard of care radiotherapy and/or before standard of care surgery.

ELIGIBILITY:
Inclusion Criteria:

* PRE-ELIGIBILITY - INCLUSION CRITERIA:
* Age >= 18 years
* Histological confirmation of newly diagnosed soft tissue sarcoma or recurrent soft tissue sarcoma >= 1-year post-treatment
* Tumors > 1 cm in diameter in largest dimension located midline within the torso or neck, retroperitoneal, or lower extremities
* Operable sarcoma, planning to receive surgery with or without neoadjuvant RT/chemotherapy at Mayo Clinic Florida. Systemic therapy is allowed during radiotherapy
* Provide informed written consent
* Willingness to participate in mandatory imaging studies at Mayo Clinic Florida

Exclusion Criteria:

* POST-ELIGIBILITY - EXCLUSION CRITERIA:
* 18F-DOPA PET uptake deemed as unacceptable for quantitative assessment
* Unable to undergo an 18F-DOPA PET/MRI scan due to standard MRI restrictions, such as for those with certain implanted devices, those who cannot fit inside the bore, or those with severe claustrophobia
* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients planning to receive surgery for high-grade soft tissue sarcoma.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2024-07-09 (Actual); Study Completion 2024-07-09 (Actual)

PRIMARY OUTCOMES:
Fluorodopa F 18 (18F-DOPA) positron emission tomography (PET) | Post-radiation therapy (RT), up to 28 days
  Correlated with pathologic response. The correlation between imaging measures and pathologic response will be evaluated using a logistic regression model for each one of the four imaging modalities separately. For each subject, 12-18 measures will be taken, and therefore, an exchangeable correlation structure will be used to model the correlation among the measures from the same patient. Giving the exploratory nature of the study, will not adjust for the multiple comparisons. Pathologic responses and imaging measurements will be summarized using point estimates, and 95% confidence interval as well, for each of the four imaging modalities.
Change in 18F-DOPA PET activity | Pre- to post-RT, up to 28 days
  Pre-radiation therapy and post-radiation therapy 18F-DOPA PET activity will be correlated with pathologic response. The correlation between imaging measures and pathologic response will be evaluated using a logistic regression model for each one of the four imaging modalities separately. For each subject, 12-18 measures will be taken, and therefore, an exchangeable correlation structure will be used to model the correlation among the measures from the same patient. Giving the exploratory nature of the study, will not adjust for the multiple comparisons. Pathologic responses and imaging measurements will be summarized using point estimates, and 95% confidence interval as well, for each of the four imaging modalities.

OTHER OUTCOMES:
Pathologic response | Through study completion, an average of 1 year
  Pathologic evaluation of resected specimens by an expert pathologist will be the gold standard for tumor diagnosis and treatment response assessment in this study. Following definitive surgery, the tumor should be examined to determine pathologic response. Since the effect of the preoperative RT may not be uniform throughout the tumor, adequate sampling is required to grade the pathologic response accurately. Tumor's pathologic response will be performed utilizing the grading system below as a guideline: grade I is defined as the percentage of necrosis less than 50%, grade II is defined as the 50%-89% necrosis in the sample, grade III is defined as 90% - 99% necrosis and grade IV is defined as 100% necrosis. The pathological endpoint is defined as the indicator of whether the percentage of necrosis is > 90%.
Imaging Endpoint Standardized uptake value (SUV) mean | Up to 3 years
  Imaging endpoints include SUV uptake value mean characteristic. Five patients will be enrolled before RT for additional PET scan for comparison of pre-RT and post-RT SUV metrics, correlated with pathology after surgery, for evaluation of 18F-DOPA PET as a marker for response assessment.
Imaging Endpoint SUV maximum | Up to 3 years
  Imaging endpoints include SUV maximum characteristic. Five patients will be enrolled before RT for additional PET scan for comparison of pre-RT and post-RT SUV metrics, correlated with pathology after surgery, for evaluation of 18F-DOPA PET as a marker for response assessment.
Imaging Endpoint Tumor-to-normal SUV | Up to 3 years
  Imaging endpoints include tumor to normal SUV characteristic. Five patients will be enrolled before RT for additional PET scan for comparison of pre-RT and post-RT SUV metrics, correlated with pathology after surgery, for evaluation of 18F-DOPA PET as a marker for response assessment.
Imaging Endpoint Total metabolic tumor volume | Up to 3 years
  Imaging endpoints include total metabolic tumor volume characteristic. Five patients will be enrolled before RT for additional PET scan for comparison of pre-RT and post-RT SUV metrics, correlated with pathology after surgery, for evaluation of 18F-DOPA PET as a marker for response assessment.
Imaging Endpoint Total tumor glycolysis | Up to 3 years
  Imaging endpoints include total tumor glycolysis characteristic. Five patients will be enrolled before RT for additional PET scan for comparison of pre-RT and post-RT SUV metrics, correlated with pathology after surgery, for evaluation of 18F-DOPA PET as a marker for response assessment.
Imaging Endpoint Tumor histogram characteristics | Up to 3 years
  Imaging endpoints include tumor histogram characteristic. Five patients will be enrolled before RT for additional PET scan for comparison of pre-RT and post-RT SUV metrics, correlated with pathology after surgery, for evaluation of 18F-DOPA PET as a marker for response assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Deanna Hasenauer, Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials